CLINICAL TRIAL: NCT05713214
Title: Long-term Follow-up After Adoptive Transfer of Genetically Modified Cell Products
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LONGENE
Record Dates: First submitted 2023-01-17; First posted 2023-02-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Relapsed Hematologic Malignancy; Refractory Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample procurement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Human gene therapy products are designed to achieve therapeutic effect through genetic modifications of human cells using retroviral or lentiviral vectors, resulting in permanent or long-acting changes in the human body. With this genetic modification comes risk of undesirable adverse events. Due to this risk, the Food and Drug Administration (FDA) and the Center for Biologics Evaluation and research (CBER) require long-term follow-up (15 years) of participants that receive investigational gene therapy products that meet defined criteria. This protocol will provide a mechanism by which to appropriately monitor participants that have received a genetically modified cellular product on a St. Jude initiated study.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, non-therapeutic study which includes routine assessment for long-term effects, as per FDA guidelines, after receipt of a gene therapy product on a St. Jude investigator-initiated clinical trial. There will be no group assignment, no use of placebo groups and no use of control subjects. Participants will enroll on this long-term follow-up study after completion of necessary follow-ups on the interventional clinical trial on which they received treatment with a genetically modified product, to complete a total of 15 years of follow-up post infusion.

Assessments will include routine history, physical exam and blood sample procurement, in accordance with FDA guidance, for 15 years post infusion of the gene therapy product. Study evaluations may be performed by a local provider in conjunction with the St. Jude research team. In addition, standard clinical data related to the subject's prior gene therapy treatment will be reviewed. The data may include, but is not limited to: patient demographics, disease history, on-going disease status updates, gene therapy product and treatment characteristics, patient clinical status, post gene therapy disease directed therapies, relapse and death

ELIGIBILITY:
Inclusion Criteria:

* Receipt of a genetically modified cell product on a St. Jude investigator-initiated study within the prior 15 years.

Exclusion Criteria:

* Inability or unwillingness of research participant and/or legal guardian/ representative to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants who have received genetically modified cell therapy products on St. Jude investigator-initiated clinical studies.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2052-12-01 (Estimated); Study Completion 2052-12-01 (Estimated)

PRIMARY OUTCOMES:
Obtain histories for detection of significant delayed medical events after receipt of a gene therapy product on a St. Jude investigator-initiated clinical trial. | 30 years
  Obtain histories for detection of significant delayed medical events after receipt of a gene therapy product on a St. Jude investigator-initiated clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Talleur, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States